CLINICAL TRIAL: NCT03548454
Title: Comparing Effectiveness of Duloxetine and Desipramine in Patients With Chronic Pain: A Pragmatic Trial Using Point of Care Randomization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vafi Salmasi, Clinical Instructor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 44758
Record Dates: First submitted 2018-04-17; First posted 2018-06-07 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Duloxetine Hydrochloride; Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Duloxetine (Experimental): Duloxetine starting at 20 mg per day and increasing to 60 mg per day as tolerated.
  Interventions: Drug: Duloxetine
- Desipramine (Experimental): Desipramine starting at 25 mg per day and increasing to 75 mg per day as tolerated.
  Interventions: Drug: Desipramine

INTERVENTIONS:
Drug: Duloxetine — Open label prescription
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Desipramine — Open label prescription
  Other Names: Norpramin
  Arms: Desipramine

SUMMARY:
Over 100 million Americans suffer from chronic pain resulting in annual cost of roughly $635 billion. Limited treatments are available for this widespread disease. The data supporting these treatments lack generalizability to patients with more serious medical and psychological comorbidities who are often excluded from explanatory efficacy trials. Our work aims to integrate randomized comparative effectiveness research with patient care. The investigators will randomize the patients and collect data using an open-source learning healthcare system already in use in our department to monitor patients' progress: Collaborative Health Outcomes Information Registry (CHOIR). Collaborative Health Outcomes Information Registry uses the National Institute of Health Patient Reported Outcomes Measurement Information System item banks for comparative metrics through computer adaptive testing. The investigators will leverage the advantage of this novel system to compare effectiveness of duloxetine and desipramine in decreasing pain in patients with chronic pain. The investigators will also compare adherence of patients to these two commonly used medications over a period of six months. This will evaluate feasibility of integrating randomized comparative effectiveness research with patient care in subspecialty clinics. Collaborative Health Outcomes Information Registry can then be applied for numerous future trials to advance our knowledge in perioperative and pain medicine.

ELIGIBILITY:
Inclusion criteria:

1. Age of 18 years old or above
2. Persistent pain for more than 3 months
3. Candidate for treatment by anti-depressant based on treating pain provider

Exclusion criteria:

1. Prior failure of duloxetine and/or desipramine (patients who have failed other TCAs or SNRIs can be considered for the trial based on the reason for previous medication failure)
2. Contraindication to taking duloxetine or desipramine
3. Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vafi Salmasi, MD., Principal Investigator — Stanford University
Locations (1):
- Stanford Pain Management Center, Redwood City, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were equally randomized to duloxetine and desipramine (43 in each arm); however, five patients chose not to take desipramine and crossed over to the duloxetine group before starting study medication.
Period: Overall Study
Arm/Group | Desipramine | Duloxetine
Started | 38 | 48
Completed | 38 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desipramine | Duloxetine | Total
Number analyzed (Participants) | 38 | 48 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.78 (14.36) | 47.25 (16.67) | 47.48 (15.62)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants with non-missing data
  Participants
    Female | 18 | 29 | 47
    Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 29 | 31 | 60
  Unknown or Not Reported | 2 | 9 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 3 | 9
  Black or African American | 1 | 0 | 1
  Unknown/Refused | 2 | 9 | 11
  White | 18 | 26 | 44
  Other | 10 | 10 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 48 | 86

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Percent of participants in each arm that had more than 30% reduction in pain intensity. Participants rated their pain on an 11-point scale (0 to 10; 0 = no pain, 10 = worst pain imaginable).
Time Frame: baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Desipramine | Duloxetine
Number analyzed (Participants) | 38 | 48
Participants | 11 | 29

2. Secondary Outcome: Physical Function
Description: National Institute of Health Patient Reported Outcomes Measurement Information System Standardized score for physical function. Raw scores were converted to T-scores with a population mean of 50 with standard deviation of 10. Overall score range: 0 to 100, higher scores correspond to better function.
Time Frame: Baseline and 6 months
Population: Participants with data at the respective time point
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Desipramine | Duloxetine
Number analyzed (Participants) | 38 | 48
T-score
  Baseline | 39.29 (7.63) | 39.07 (6.33)
  6-month: number analyzed (Participants) | 36 | 45
  6-month | 41.9 (8.91) | 39.39 (6.98)
  Change from baseline at 6-month: number analyzed (Participants) | 36 | 45
  Change from baseline at 6-month | 2.54 (5.83) | 1.36 (3.88)

3. Secondary Outcome: Pain Interference
Description: National Institute of Health Patient Reported Outcomes Measurement Information System Standardized score for pain interference. Raw scores were converted to T-scores with a population mean of 50 with standard deviation of 10. Overall score range: 0 to 100, higher scores correspond to worse pain interference.
Time Frame: Baseline and 6 months
Population: Participants with data at the respective time point
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Desipramine | Duloxetine
Number analyzed (Participants) | 38 | 48
T-score
  Baseline | 64.37 (7.1) | 64.93 (6.48)
  6-month: number analyzed (Participants) | 36 | 45
  6-month | 60.82 (7.1) | 62.11 (6.98)
  Change from baseline at 6-month: number analyzed (Participants) | 36 | 45
  Change from baseline at 6-month | -4.29 (7.57) | -4.06 (7.51)

4. Secondary Outcome: Depression
Description: National Institute of Health Patient Reported Outcomes Measurement Information System Standardized score for depression. Raw scores were converted to T-scores with a population mean of 50 with standard deviation of 10. Overall score range: 0 to 100, higher scores correspond to more severe depression.
Time Frame: Baseline and 6 months
Population: Participants with data at the respective time point
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Desipramine | Duloxetine
Number analyzed (Participants) | 38 | 48
T-score
  Baseline | 52.98 (9.40) | 54.24 (8.89)
  6-month: number analyzed (Participants) | 36 | 45
  6-month | 52.54 (9.7) | 53.39 (11.93)
  Change from baseline at 6-month: number analyzed (Participants) | 36 | 45
  Change from baseline at 6-month | -3.24 (6.58) | -1.14 (12.83)

5. Secondary Outcome: Anxiety
Description: National Institute of Health Patient Reported Outcomes Measurement Information System Standardized score for anxiety. Raw scores were converted to T-scores with a population mean of 50 with standard deviation of 10. Overall score range: 0 to 100, higher scores correspond to more severe anxiety.
Time Frame: Baseline and 6 months
Population: Participants with data at the respective time point
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Desipramine | Duloxetine
Number analyzed (Participants) | 38 | 48
T-score
  Baseline | 54.39 (10.21) | 54.65 (8.99)
  6-month: number analyzed (Participants) | 36 | 45
  6-month | 54.97 (9.65) | 54.01 (11.72)
  Change from baseline at 6-month: number analyzed (Participants) | 36 | 45
  Change from baseline at 6-month | -1.2 (7.11) | -1.29 (11.89)

6. Secondary Outcome: Adherence
Description: Number of participants who completed 6-month therapy based on prescription records.
Time Frame: Monthly for 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Desipramine | Duloxetine
Number analyzed (Participants) | 38 | 48
Participants | 18 | 24

ADVERSE EVENTS:
Time Frame: During 6 months duration of the study
Description: All participants were systematically inquired about presence of adverse events during each study survey
Arm/Group | Desipramine | Duloxetine
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/48
Other Adverse Events (participants affected / at risk) | 6/38 | 4/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desipramine (N=38) | Duloxetine (N=48)
Did not tolerate (Investigations) | 1 (1) | 0 (0) — Patient mentioned they did not tolerate the medication and refused to provide more information why
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0) — Daytime drowsiness
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — prolonged bleeding and easier bruising
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) — urinary frequency and urgency
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Increased pain (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT03548454/Prot_001.pdf
  • Statistical Analysis Plan: Original Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT03548454/SAP_002.pdf
  • Statistical Analysis Plan: Revised Statistical Analysis Plan (2025-03-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT03548454/SAP_003.pdf